CLINICAL TRIAL: NCT07283718
Title: The Association Between Axillary Lymph Node Metastasis Patterns and Breast Cancer Prognosis：a Real-world Study
Brief Title: The Association Between Axillary Lymph Node Metastasis Patterns and Breast Cancer Prognosis
Status: Active, not recruiting | Type: Observational
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: LY2025-298-B
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALND: breast cancer patients receiving axillary lymph mode dissection
  Interventions: Procedure: ALND

INTERVENTIONS:
Procedure: ALND — axillary lymph node dissection

SUMMARY:
This is a real-world multicentre study to investigate the metastatic pattern of axillary lymph node and its association with breast cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathologically confirmed invasive primary breast cancer

Exclusion Criteria:

* De novo stage IV breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were pathologically diagnosed primary invasive breast cancer from October 2013 to December 2023. They had axillary lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 2467 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the date of ALND until time of event up to 3 years
  Disease-free survival time is defined as the time from the date of axillary lymph node dissection until the date of the first occurrence of local/regional relapse, distant recurrence, contralateral breast cancer, second malignancy and death from any cause.

SECONDARY OUTCOMES:
Recurrence-free survival | From the date of ALND until time of event up to 3 years
  Recurrence-free survival time is defined as the time from the date of axillary lymph node dissection until the date of the first occurrence of local/regional recurrence, distant recurrence and death from any cause
Overall survival | From the date of ALND until time of event up to 3 years
  Overall survival time is defined as the time from the date of axillary lymph node dissection until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China